CLINICAL TRIAL: NCT00855517
Title: A Partially Masked, Phase 2 Study of the Latanoprost Punctal Plug Delivery System (L-PPDS) in Subjects With Ocular Hypertension (OH) or Open-Angle Glaucoma (OAG)
Brief Title: A Phase 2 Study of the Latanoprost Punctal Plug Delivery System in Subjects With Ocular Hypertension or Open-Angle Glaucoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPL GLAU 06
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Punctal Plug (Experimental)
  Interventions: Drug: Latanoprost-PPDS

INTERVENTIONS:
Drug: Latanoprost-PPDS — Control of IOP compared to baseline for the experimental dose of Latanoprost-PPDS for 6 weeks or until loss of efficacy.

SUMMARY:
The purpose of this study is to evaluate IOP response to experimental dose of Latanoprost- PPDS in subjects with ocular hypertension or open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 yrs of age with ocular hypertension or open-angle glaucoma
* Subjects who have a best corrected visual acuity of 20/100 or better

Exclusion Criteria:

* Subjects who wear contact lenses.
* Uncontrolled medical conditions
* Subjects requiring chronic topical artifical tears, lubricants and/or requiring any other chronic topical medications
* Subjects who have a history of chronic or recurrent inflammatory eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
IOP change from baseline | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Cuzzani, MD, Study Director — QLT Inc.